CLINICAL TRIAL: NCT05915351
Title: A Phase II Open-Label Study of Enfortumab Vedotin in Patients With Previously Treated Locally Advanced, Recurrent, or Metastatic Pancreatic Adenocarcinoma (EPIC)
Brief Title: Enfortumab Vedotin in Previously Treated Locally Advanced or Metastatic Pancreatic Cancer (EPIC)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Anup Kasi, MD, MPH, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00150104
Record Dates: First submitted 2023-05-23; First posted 2023-06-23 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Pancreas Adenocarcinoma; Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — enfortumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Experimental): Enfortumab vedotin, 1.25 mg/kg IV on D 1,8,15 every 28 days
  Interventions: Drug: Enfortumab vedotin

INTERVENTIONS:
Drug: Enfortumab vedotin — Enfortumab vedotin 1.25 mg/kg on D1, D8, D15 every 28 days
  Other Names: Padcev

SUMMARY:
A Phase II Open-Label Study of Enfortumab Vedotin in Patients with Previously Treated Locally Advanced, Recurrent, or Metastatic Pancreatic Adenocarcinoma (EPIC)

DETAILED DESCRIPTION:
Enfortumab vedotin is an antibody-drug conjugate that delivers the microtubule-disrupting agent monomethyl auristatin E (MMAE) to cells expressing Nectin-4. Enfortumab vedotin is FDA approved for bladder cancer.

This is a phase II, open-label, study to evaluate the efficacy, safety and tolerability of Enfortumab vedotin in participants with previously treated locally advanced, recurrent, or metastatic pancreatic adenocarcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Ability of participant OR Legally Authorized Representative (LAR) to understand this study, and participant or LAR willingness to sign a written informed consent
2. Males and females age ≥ 18 years
3. Subjects with locally advanced, recurrent or metastatic pancreatic adenocarcinoma after progressing or intolerant to at least one line of systemic therapy
4. ECOG Performance Status 0 - 1 (Appendix A.)
5. Measurable disease by RECIST 1.1
6. Women of childbearing potential must have a negative urine or serum pregnancy test 7 days prior to initiating treatment.
7. Adequate archival tissue from prior biopsy for biomarker evaluation or willingness to undergo tissue biopsy before treatment starts and on treatment. Patients who, in the opinion of the investigator, do not have tissue that can be safely biopsied are excepted.
8. Absolute Neutrophil Count >1.5K/UL NOTE: Patients with established diagnosis of benign neutropenia are eligible to participate with ANC between 1000-1500 if in the opinion of treating physician the trial treatment does not pose excessive risk of infection to the patient.
9. Platelets >100K/UL
10. Hemoglobin ≥ 9 g/dL
11. Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 50 mL/min using the Cockcroft-Gault equation
12. Total bilirubin ≤ 1.5 x ULN OR direct bilirubin ≤ 1 x ULN
13. Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x ULN unless liver metastases are present, in which case they must be ≤ 5 x ULN
14. Women of child-bearing potential and men with partners of child-bearing potential must agree to practice sexual abstinence or to use the forms of contraception listed in Child-Bearing Potential/Pregnancy section for the duration of study participation and

    * Females: at least 2 months after the last dose of the study medication.
    * Males: at least 4 months after the last dose of the study medication.

Exclusion Criteria:

1. Simultaneously enrolled in any therapeutic clinical trial
2. Current or anticipating use of other anti-neoplastic or investigational agents while participating in this study
3. Diagnosed with a psychiatric illness or is in a social situation that would limit compliance with study requirements
4. Has a known allergic reaction to any excipient contained in the study drug formulation
5. Active Grade 3 (per the NCI CTCAE, Version 5.0) or higher viral, bacterial, or fungal infection within 2 weeks prior to the first dose of study treatment.
6. Ongoing sensory or motor neuropathy Grade 2 or higher.
7. Active central nervous system (CNS) metastases. Patients with treated CNS metastases are permitted on study if all the following are true:

   1. CNS metastases have been clinically stable for at least 6 weeks prior to screening and baseline scans show no evidence of new or enlarged metastasis.
   2. If requiring steroid treatment for CNS metastases, the patient is on a stable dose <10 mg/day of prednisone or equivalent for at least 2 weeks.
   3. Patient does not have leptomeningeal disease
8. Patients with conditions requiring high doses of steroids (>10 mg/day of prednisone or equivalent) or other immunosuppressive medications are excluded. Inhaled or topical steroids are permitted in the absence of active autoimmune disease.
9. Prior treatment with enfortumab vedotin or other MMAE-based antibody-drug conjugates (ADCs).
10. Currently receiving systemic antimicrobial treatment for active infection (viral, bacterial, or fungal) at the time of first dose of enfortumab vedotin. Routine antimicrobial prophylaxis is permitted.
11. Patients with a positive hepatitis B surface antigen and/or antihepatitis B core antibody; patients with a negative polymerase chain reaction (PCR) assay are permitted with either universal prophylaxis or the use of a pre-emptive approach.
12. Active hepatitis C infection or known human immunodeficiency virus (HIV) infection NOTE: Patients who have been curatively treated for hepatitis C infection are permitted if they have documented sustained virologic response of 12 weeks. No HIV testing is required unless mandated by local health authority.
13. Patients with active tuberculosis based on medical history.
14. Documented history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms (including congestive heart failure) consistent with NYHA Class III-IV within 6 months prior to the first dose of enfortumab vedotin.
15. Radiotherapy or major surgery within 2 weeks prior to first dose of study drug. Patient must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
16. Patients with active keratitis or corneal ulcerations. Patients with superficial punctate keratitis are allowed if the disorder is being adequately treated in the opinion of the investigator.
17. History of idiopathic pulmonary fibrosis; organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
18. Prior allogeneic stem cell or solid organ transplant.
19. Administration of a live, attenuated vaccine within 30 days prior to first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, BCG, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
20. Other underlying medical condition that, in the opinion of the investigator, would impair the ability of the patient to receive or tolerate the planned treatment and follow-up; any known psychiatric or substance abuse disorders that would interfere with cooperating with the requirements of the study.
21. Patients with uncontrolled diabetes. Uncontrolled diabetes is defined as hemoglobin A1c (HbA1c) ≥8% or HbA1c 7% to <8% with associated diabetes symptoms (polyuria or polydipsia) that are not otherwise explained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Every 8 weeks until disease progression or end of study (approximately 2 years), whichever is earlier
  To determine anti-tumor activity by overall response rate (ORR) using RECIST 1.1

SECONDARY OUTCOMES:
Safety and Tolerability | Adverse Event Collection and Review will occur on Days 1,8,15 for each 28-day cycle until disease progression or end of treatment (approximately 2 years)
  To determine treatment safety based on toxicities evaluated according to National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 in patients who have received at least one dose of enfortumab vedotin
Duration of Response (DOR) | approximately 2 years
  To determine anti-tumor activity by duration of response (DOR)
Disease Control Rate (DCR) | approximately 2 years
  To determine anti-tumor activity by disease control rate (DCR)
Progression Free Survival (PFS) | Every 8 weeks until disease progression or subsequent therapy assessed up to 2 years
  To determine progression free survival (PFS)
Overall Survival (OS) | Every 3 months for 12 months after End of Treatment
  To determine overall survival (OS)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Cancer Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No